CLINICAL TRIAL: NCT00490477
Title: Polymyxin-B Hemoperfusion Inactivates Circulating Proapoptotic Factors
Brief Title: The Effects of Polymyxin-B Protects on Sepsis Induced Kidney Dysfunction: a Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: V. M. Ranieri, MD, University of Turin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N-257
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Results first posted 2010-06-04 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Gram-Negative Bacterial Infections; Sepsis
Keywords: acute renal failure; lipopolysaccharide; tubular apoptosis; Polymyxin-B fiber; Severe sepsis from gram negative infection
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Sepsis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONVENTIONAL (No Intervention)
- POLYMYXIN-B (Active Comparator): an extracorporeal LPS removal
  Interventions: Device: Polymyxin -B fiber hemoperfusion system

INTERVENTIONS:
Device: Polymyxin -B fiber hemoperfusion system — two hours treatment for two days
  Other Names: PMX-B
  Arms: POLYMYXIN-B

SUMMARY:
Aim of the study is to verify whether Polymyxin-B hemoperfusion protects from renal dysfunction in patients with severe sepsis from gram negative infection.

DETAILED DESCRIPTION:
Acute renal failure (ARF) is a frequent complication in sepsis, in nearly to 50% of the cases, and the mortality rate is higher, compare to patients with ARF alone (70% vs 45%). Clinical and experimental studies demonstrated the key role of apoptosis, or programmed cell death, in the induction of tubular and glomerular injury in the course of sepsis. Indeed, it has been shown that inflammatory cytokines and lipopolysaccharide (LPS) cause renal tubular cell apoptosis via Fas- and caspase-mediated pathways. In addition, LPS is able to alter the normal expression pattern of sodium, urea and glucose renal transporters and to modulate tubular polarity by changing the expression of tight junction proteins with consequent back-leakage of tubular fluid in the interstitial spaces and enhancement of the inflammatory process. Therefore a novel extracorporeal therapy to remove circulating LPS, using the Polymyxin-B fiber (PMX-B) cartridge was developed. The PMX-B cartridge is an extracorporeal hemoperfusion device and consists of a polystyrene-based, fibrous adsorbent on which the polymyxin B antibiotic is covalently immobilized as a ligand to adsorb endotoxin.

Aim of this study is to verify whether the removal of LPS, using the PMX-B hemoperfusion system, protects from acute renal failure, reduces the need for Renal Replacement Therapy (RRT) and consequently improves the outcome in severe sepsis from gram negative infection.

ELIGIBILITY:
Inclusion Criteria:

* Endotoxemia associated to severe sepsis

Exclusion Criteria:

* Age < 18 years old
* Organ transplantation
* Hemorrhagic shock
* Thrombophilia
* Chronic renal failure
* Cardiogenic shock
* APACHE II score > 30
* Lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-05; Primary Completion 2007-07 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: marco ranieri, MD, Study Director — University of Turin, Department of Anesthesia and Intensive Care Medicine; marco ranieri, MD, Principal Investigator — University of Turin, Department of Anesthesia and Intensive Care Medicine
Locations (1):
- University of Turin, Department of anesthesia and Intensive Care Medicine, Turin, Italy

REFERENCES:
- [Result] Cantaluppi V, Assenzio B, Pasero D, Romanazzi GM, Pacitti A, Lanfranco G, Puntorieri V, Martin EL, Mascia L, Monti G, Casella G, Segoloni GP, Camussi G, Ranieri VM. Polymyxin-B hemoperfusion inactivates circulating proapoptotic factors. Intensive Care Med. 2008 Sep;34(9):1638-45. doi: 10.1007/s00134-008-1124-6. Epub 2008 May 8. PMID 18463848

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Treatment (CONV): patients with Gram-negative severe sepsis who received standard care according to Surviving Sepsis Campaign guidelines
- Polymyxin-B Hemoperfusion Treatment (PMX-B): patients with Gram-negative severe sepsis treated with standard therapy, according to the Surviving Sepsis Campaign, and an extracorporeal therapy with a PMX-B filter that could remove LPS
Period: Overall Study
Arm/Group | Conventional Treatment (CONV) | Polymyxin-B Hemoperfusion Treatment (PMX-B)
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Treatment (CONV) | Polymyxin-B Hemoperfusion Treatment (PMX-B) | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 2 | 4 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 61 (10) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Italy | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Not Requiring Renal Replacement Therapy (RRT)
Time Frame: 28 days from the admission
Measure: Number; unit: participants
Arm/Group | Conventional Treatment (CONV) | Polymyxin-B Hemoperfusion Treatment (PMX-B)
Number analyzed (Participants) | 8 | 8
participants | 3 | 1

2. Secondary Outcome: The Reduction of the Number of Apoptotic Cells, Stimulated With Plasma Derives From Septic Patients With Gram Negative Infection, Treated With PMX-B Hemoperfusion, on Immortalized Tubular and Glomerular Cell Cultures.
Time Frame: 72 hours after randomization
Reporting Status: Not Posted, anticipated posting 2007-04
Measure: Number; unit: cells

ADVERSE EVENTS:
Arm/Group | Conventional Treatment (CONV) | Polymyxin-B Hemoperfusion Treatment (PMX-B)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No